CLINICAL TRIAL: NCT04770636
Title: Glucose Disturbances in the First Day of Life in Preterm Infants and Health-related Quality of Life: is There a Correlation?
Brief Title: Glucose Disturbances in Premature Infants and Quality of Life
Status: Enrolling by invitation | Type: Observational
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Kristina Lah Tomulić, MD, PhD, Clinical Hospital Center Rijeka
Other Study IDs: KBC-ped-endo
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Neonatal Hypoglycemia; Neonatal Hyperglycaemia
Keywords: Preterm birth, Hypoglycemia, Hyperglycemia, Quality of life
MeSH Terms: conditions — Premature Birth; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the correlation between preterm birth, glucose level in the first two hours of life and health related quality of life in the age of 8 months and 7 years

DETAILED DESCRIPTION:
All premature infants treated from August 2013-August 2014 in two Neonatal intensive care units (NICUs) are included in this study. Glucose levels was analyzed two hours after birth. In the age of 8 months parents completed the questionnaire Pediatric Quality of Life - Infant scale. The questionnaire Quality of life for children 5-7 years and for their parents will be offered to them in the next 4 months.

We will investigate if there is a correlation between glucose levels and quality of life in premature infants, and if quality of life changes over years.

ELIGIBILITY:
Inclusion Criteria: All premature infants treated in two neonatal intensive units in Clinical Hospital centre Rijeka in the year 2013.- 2014. To reach to final outcome, all questionnaires must be completed.

-

Exclusion Criteria: All deceased premature children born in the study period.

-

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants are all premature infants (born before 37th gestational week) treated in two intensive care units: Neonatal intensive unit cares for inborn premature infants and Pediatric intensive care unit takes care for premature infant born in other hospitals in three counties.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-08-01 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of glucose levels in prematures after birth and Quality of life in the age of 7 years | 7 years
  Glucose level was measured two hours after birth in all premature infants. In the age of 8 months and 7 years Quality of life was measured using the questionnaire Paediatric Quality of Life (PedsQL) - Infant scale (6-12 months). The PedsQL Young Child report (5-7 years) and Parent report for Young children (5-7 years) will be offered to one parent/caregiver. In both scales minimum value is zero and maximum is 100; Higher score means better quality of life. The correlation between glucose levels in premature infants and quality of life will be investigated.

SECONDARY OUTCOMES:
Comparison of Quality of life in premature infants in the age of 8 months and 7 years | 6,5 years
  The questionnaire Paediatric Quality of Life (PedsQL) - Infant scale (6-12 months) was completed by a parent/caregiver of premature infants in the age of 8 months. In the age of 7 years the questionnaire PedsQL Young Child report (5-7 years) and Parent report for Young children (5-7 years) will be offered to parents/caregivers. The quality of life will be compared in these two intervals to investigate the changes in quality of life over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre, Rijeka, Primorsko-goranska County, Croatia